CLINICAL TRIAL: NCT04292899
Title: A Phase 3 Randomized Study to Evaluate the Safety and Antiviral Activity of Remdesivir (GS-5734™) in Participants With Severe COVID-19
Brief Title: Study to Evaluate the Safety and Antiviral Activity of Remdesivir (GS-5734™) in Participants With Severe Coronavirus Disease (COVID-19)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-540-5773; 2020-000841-15 (EudraCT Number); ISRCTN15874265 (Other: ISRCTN)
Expanded Access: NCT04323761 (Approved for marketing)
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Remdesivir (RDV), 5 Days (Experimental): Participants will receive continued standard of care therapy together with RDV 200 mg on Day 1 followed by RDV 100 mg on Days 2, 3, 4, and 5.
  Interventions: Drug: Remdesivir; Drug: Standard of Care
- Part A: Remdesivir, 10 Days (Experimental): Participants will receive continued standard of care therapy together with RDV 200 mg on Day 1 followed by RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10.
  Interventions: Drug: Remdesivir; Drug: Standard of Care
- Part B: Remdesivir, 10 Days (Extension) (Experimental): Part B (Extension) will enroll participants after enrollment to Part A is complete. Participants will receive continued standard of care therapy together with RDV 200 mg on Day 1 followed by RDV 100 mg on Days 2-10.
  Interventions: Drug: Remdesivir; Drug: Standard of Care
- Part B: Remdesivir 10 days (Mechanically Ventilated) (Experimental): Participants on mechanical ventilation will receive continued standard of care therapy together with RDV 200 mg on Day 1 followed by RDV 100 mg on Days 2-10
  Interventions: Drug: Remdesivir; Drug: Standard of Care

INTERVENTIONS:
Drug: Remdesivir — Administered as an intravenous infusion
  Other Names: GS-5734™; Veklury®
Drug: Standard of Care — Standard of Care Treatment for COVID-19 Infection

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 2 remdesivir (RDV) regimens with respect to clinical status assessed by a 7-point ordinal scale on Day 14.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent, or enrolled under International Conference on Harmonization (ICH) E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (age ≥ 18), or willing and able to provide assent (age ≥ 12 to < 18, where locally and nationally approved) prior to performing study procedures
* Aged ≥ 18 years (at all sites), or aged ≥ 12 and < 18 years of age weighing ≥ 40 kg (where permitted according to local law and approved nationally and by the relevant institutional review board (IRB) or independent ethics committee (IEC))
* Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR) test ≤ 4 days before randomization
* Currently hospitalized
* Peripheral capillary oxygen saturation (SpO2) ≤ 94% or requiring supplemental oxygen at screening

Key Exclusion Criteria:

* Participation in any other clinical trial of an experimental treatment for COVID-19
* Concurrent treatment with other agents with actual or possible direct acting antiviral activity against SARS-CoV-2 is prohibited < 24 hours prior to study drug dosing
* Evidence of multiorgan failure
* Mechanically ventilated [including veno-venous (V-V) extracorporeal membrane oxygenation (ECMO)] ≥ 5 days, or any duration of veno-arterial (V-A) ECMO.
* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 X upper limit of normal (ULN)
* Creatinine clearance < 50 mL/min using the Cockcroft-Gault formula for participants ≥ 18 years of age {Cockcroft 1976} and Schwartz Formula for participants < 18 years of age

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4891 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (182):
- United States (106):
  - Kaiser Permanente Los Angeles Medical Center, 3340 E. La Palma Avenue, Anaheim, California
  - Alta Bates Summit Medical Center, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Eden Medical Center, Castro Valley, California
  - Kaiser Permanente Los Angeles Medical Center, 9333 Imperial Highway, Downey, California
  - Kaiser Permanente Los Angeles Medical Center, 9961 Sierra Ave, Fontana, California
  - St Joseph Hospital Eureka, Fortuna, California
  - Kaiser Permanente Los Angeles Medical Center, 25825 S. Vermont Ave., Harbor City, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, 6041 Cadillac Ave., Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, 5601 De Soto Avenue, Los Angeles, California
  - Mission Hospital Regional Medical Center, Mission Viejo, California
  - Kaiser Permanente Los Angeles Medical Center, 27300 Iris Avenue, Moreno Valley, California
  - El Camino Hospital, Mountain View, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Kaiser Permanente Los Angeles Medical Center, 2295 S. Vineyard Avenue, Ontario, California
  - The Center for Cancer Prevention and Treatment at St. Joseph Hospital of Orange, Orange, California
  - Kaiser Permanente Los Angeles Medical Center, 13651 Willard Street, Panorama City, California
  - Kaiser Permanente Los Angeles Medical Center, 10800 Magnolia Avenue, Riverside, California
  - Sutter Medical Center Sacramento, One Medical Plaza, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente Los Angeles Medical Center, 4647 Zion Avenue, San Diego, California
  - Kaiser Permanente Los Angeles Medical Center, 9455 Clairemont Mesa Blvd, San Diego, California
  - Kaiser Permanente Oakland Medical Center, 1200 El Camino Real, San Francisco, California
  - California Pacific Medical Center-Infectious Disease Associates Medical Group, San Francisco, California
  - Kaiser Permanente Oakland Medical Center, 2425 Geary Blvd, San Francisco, California
  - Kaiser Permanente Oakland Medical Center, 250 Hospital Parkway, Suite 850, San Jose, California
  - Kaiser Permanente Oakland Medical Center, 2500 Merced St, San Leandro, California
  - Kaiser Permanente Oakland Medical Center, 700 Lawrence Expressway, Santa Clara, California
  - Providence St. Johns Medical Center, Santa Monica, California
  - Sutter Santa Rosa Regional Hospital, Santa Rosa, California
  - Stanford Hospital, Stanford, California
  - University of Colorado Denver, University of Colorado Hospital, Aurora, Colorado
  - SCL Health St. Joseph Hospital, 1375 East 19th Ave, Denver, Colorado
  - SCL Health St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - SCL Health St. Joseph Hospital, 200 Exempla Circle., Lafayette, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Kaiser Permanente Hawaii Moanalua Medical Center, Honolulu, Hawaii
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Holy Cross Hospital, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham & Women's Hospital and Harvard Medical School, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The University of Michigan Hospitals and Health Systems, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Providence St Patrick Hospital and International Heart Institute of MT Foundation, Missoula, Montana
  - Darmouth-Hitchhock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Hillsborough, New Jersey
  - Robert Wood Johnson University Hospital Somerset, 1 RWJ Place, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, 201 Lyons Avenue, Newark, New Jersey
  - St. Joseph's University Medical Center, Paterson, New Jersey
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Danbury Hospital, Lagrangeville, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, 270-05 76th Ave, New Hyde Park, New York
  - Icahn School of Medicine at Mount Sinai, 350 East 17th Street, New York, New York
  - Icahn School of Medicine at Mount Sinai, 1000 10th Avenue, New York, New York
  - Icahn School of Medicine at Mount Sinai, 440 West 114th St., New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - James J. Peters Veterans Administration Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Kaiser Sunnyside Medical Center, 2875 NW Stucki Ave, Hillsboro, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Sunnyside Medical Center, Portland, Oregon
  - Hospital of the University of Pennsylvania, 51 N. 31st Street, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Prisma Health Richland Hospital, 701 Grove Road, Greenville, South Carolina
  - The Liver Institute of Methodist Dallas Medical Center, Dallas, Texas
  - UT Southwestern Medical Center Amelia Court, HIV Research Clinic, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center Amelia Court, HIV Research Clinic, 5201 Harry Hines Blvd., Dallas, Texas
  - UT Southwestern Medical Center Amelia Court, HIV Research Clinic, 6201 Harry Hines Blvd, Dallas, Texas
  - Baylor University Medical Center, 1400 8th Ave, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor University Medical Center, 2401 S. 31st St., Temple, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Virginia Hospital Center, Arlington, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - VCU Health Medical Center, Richmond, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Kadlec Regional Medical Center, Kennewick, Washington
  - Providence St. Peter Hospital, Olympia, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Center for Comprehensive Care, Seattle, Washington
  - MultiCare Deaconess Hospital, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - St Joseph Medical Center, Tacoma, Washington
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China
- France (5):
  - CHU Pellegrin, Bordeaux
  - CHU de Montpellier-Hopital Gui de Chauliac, Montpelier Cedex 5
  - CHU de Nantes-Hotel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - Hopital Saint Antoine, Paris
- Germany (8):
  - Charite Universitatsmedizin Berlin, Campus Virchow-Klinikum, Medizinische Klinik Infektiologie Pneumologie, Berlin
  - Universitatsklinikum Dusseldorf, Klinik fur Gastroenterologie, Hepatologie und Infektiologie, Düsseldorf
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Klinikum St. Georg gGmbH Klinik fur Infektiologie, Tropenmedizin, Nephrologie und Rheumatologie, Leipzig
  - Klinikum rechts der Isar der TU Munchen, Klinik und Poliklinik Innere Medizin 2, Munich
  - Klinik für Hämatologie, Onkologie, Immunologie, München
  - Robert-Bosch-Krankenhaus (RBK), Klinik Schillerhohe (KSH) und Dr. Margarete Fischer-Bosch-Institut fur klinische Pharmakologie (IKP), Stuttgart
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Italy (12):
  - UOC Malattie Infettive, ASST Papa Giovanni XXIII, Bergamo
  - ASST degli Spedali Civili di Brescia, Brescia
  - ASST di Cremona - Azienda Socio Sanitaria Territor, Cremona
  - UO Malattie Infettive, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - UOC Malattie Infettive, IRCCS Ospedale San Raffaele, Milan
  - Dipartimento di Malattie Infettive, Malattie Infettive I- Malattie Infettive III, AssT Fatebenefratelli Sacco Ospedale Luigi Sacco, Milan
  - UOC Medicina Di Laboratorio, Azienda Ospedaliera di Padova, Padova PD
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - UOC Malattie Infettive I, Fondazione IRCCS Policlinio San Matteo, Pavia
  - Ospedale Guglielmo da Saliceto AUSL di Piacenza, Piacenza
  - UOC Malattie Infettive ad Alta Intensita di Cure, Istituto Nazionale Malattie Infettive Lazzaro Spallanzani I.R.C.C.S., Roma
  - Clinica Universitaria Malattie Infettive, Ospedale Amedeo di Savoia, Torino
- Japan (3):
  - Yokohama Municipal Citizen's Hospital, Kanagawa
  - Nagoya City East Medical Center, Nagoya
  - Tokyo Metropolitan Bokutoh Hospital, Tokyo
- Netherlands (3):
  - Amsterdam University Medical Centre - Location AMC, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Centre, Rotterdam
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Centre for Infectious Diseases, Tan Tock Seng Hospital, Singapore
- South Korea (3):
  - Kyungpook National University Hospital, Daegu
  - Seoul Medical Center, Seoul
  - National Medical Center, Seoul
- Spain (12):
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Cruces, Bizkaia
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (3):
  - Sahlgrenska University Hospital, Ostra, Gothenburg
  - SUS (Skanes University Hospital), Malmo
  - Karolinska University Hospital, Stockholm
- Switzerland (3):
  - Hopitaux Universitaires de Genève, Geneva
  - Ospedale Regionale di Locarno La Carità, Lugano
  - Universitätsspital Zürich, Zurich
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (14):
  - Imperial College Healthcare NHS Trust, London, Greater London
  - Royal Infirmary of Edinburgh, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Royal Lancaster Hospital, Lancaster
  - Liverpool University Hospital, Liverpool
  - Northwick Park Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - King's College Hospital NHS Trust, London
  - University College London, London
  - Manchester University NHS Foundation Trust, Manchester
  - Pennine Acute Hospitals NHS Trust, Manchester
  - Derriford Hospital, Plymouth
  - Sheffield Teaching Hospitals, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Background] Goldman JD, Lye DCB, Hui DS, Marks KM, Bruno R, Montejano R, Spinner CD, Galli M, Ahn MY, Nahass RG, Chen YS, SenGupta D, Hyland RH, Osinusi AO, Cao H, Blair C, Wei X, Gaggar A, Brainard DM, Towner WJ, Munoz J, Mullane KM, Marty FM, Tashima KT, Diaz G, Subramanian A; GS-US-540-5773 Investigators. Remdesivir for 5 or 10 Days in Patients with Severe Covid-19. N Engl J Med. 2020 Nov 5;383(19):1827-1837. doi: 10.1056/NEJMoa2015301. Epub 2020 May 27. PMID 32459919
- [Derived] Fusco D, Malenica I, Gunthard HF, Gupta SK, Kurbegov D, Balani B, Olender S, Aberg JA, Telep LE, Tian Y, Blair C, Wu G, Haubrich RH, Wang CY, Chokkalingam AP, Osinusi AO, Wendtner CM, Gottlieb RL. Remdesivir for Treatment of COVID-19 Requiring Oxygen Support: A Cross-Study Comparison From 2 Large, Open-Label Studies. Clin Infect Dis. 2024 Nov 22;79(5):1182-1189. doi: 10.1093/cid/ciae336. PMID 38920297
- [Derived] Jacobson KB, Rao M, Bonilla H, Subramanian A, Hack I, Madrigal M, Singh U, Jagannathan P, Grant P. Patients With Uncomplicated Coronavirus Disease 2019 (COVID-19) Have Long-Term Persistent Symptoms and Functional Impairment Similar to Patients with Severe COVID-19: A Cautionary Tale During a Global Pandemic. Clin Infect Dis. 2021 Aug 2;73(3):e826-e829. doi: 10.1093/cid/ciab103. PMID 33624010
- [Derived] Olender SA, Perez KK, Go AS, Balani B, Price-Haywood EG, Shah NS, Wang S, Walunas TL, Swaminathan S, Slim J, Chin B, De Wit S, Ali SM, Soriano Viladomiu A, Robinson P, Gottlieb RL, Tsang TYO, Lee IH, Hu H, Haubrich RH, Chokkalingam AP, Lin L, Zhong L, Bekele BN, Mera-Giler R, Phulpin C, Edgar H, Gallant J, Diaz-Cuervo H, Smith LE, Osinusi AO, Brainard DM, Bernardino JI; GS-US-540-5773 and GS-US-540-5807 Investigators. Remdesivir for Severe Coronavirus Disease 2019 (COVID-19) Versus a Cohort Receiving Standard of Care. Clin Infect Dis. 2021 Dec 6;73(11):e4166-e4174. doi: 10.1093/cid/ciaa1041. PMID 32706859

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Europe, and Asia. The first participant was screened on 06 March 2020. The last study visit occurred on 30 June 2020.
Pre-assignment Details: 4958 participants were screened. 4891 participants were enrolled. 4 participants in Part A and 49 participants in Part B did not receive treatment and are not included in the analyses.
Groups:
- Part A: Remdesivir (RDV) for 5 Days: Participants received continued standard of care (SOC) therapy together with intravenous (IV) RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2-5.
- Part A: Remdesivir for 10 Days: Participants received continued SOC therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2-10.
- Part B: Remdesivir for 10 Days (Mechanically Ventilated Group): Participants on mechanical ventilation received continued SOC therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2-10.
- Part B: Remdesivir for 10 Days (Extension Group): Participants who were not mechanically ventilated received continued SOC therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2-10.
Period: Overall Study
Arm/Group | Part A: Remdesivir (RDV) for 5 Days | Part A: Remdesivir for 10 Days | Part B: Remdesivir for 10 Days (Mechanically Ventilated Group) | Part B: Remdesivir for 10 Days (Extension Group)
Started | 200 | 197 | 844 | 3597
Completed | 168 | 164 | 621 | 2952
Not Completed | 32 | 33 | 223 | 645
Not completed — Death | 21 | 28 | 188 | 371
Not completed — Lost to Follow-up | 8 | 4 | 22 | 235
Not completed — Withdrew consent | 1 | 0 | 11 | 32
Not completed — Adverse Event | 2 | 1 | 2 | 2
Not completed — Investigator's Discretion | 0 | 0 | 0 | 3
Not completed — Non-compliance With Study Drug | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Part A: Safety Analysis Set included participants who were randomized into part A of the study and received at least 1 dose of study treatment.
  Part B: Expanded RDV-Treated Analysis Set included participants who were enrolled into part B of the study and received at least 1 dose of study treatment.
Groups:
- Part A: Remdesivir (RDV) for 5 Days: Participants received continued SOC therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2-5.
- Total: Total of all reporting groups
Arm/Group | Part A: Remdesivir (RDV) for 5 Days | Part A: Remdesivir for 10 Days | Part B: Remdesivir for 10 Days (Mechanically Ventilated Group) | Part B: Remdesivir for 10 Days (Extension Group) | Total
Number analyzed (Participants) | 200 | 197 | 844 | 3597 | 4838
Age, Customized [Count of Participants; unit: Participants]
  Age Categories: < 65 | 116 | 113 | 581 | 2399 | 3209
  Age Categories: ≥ 65 | 84 | 84 | 263 | 1198 | 1629
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 64 | 312 | 1351 | 1807
  Male | 120 | 133 | 532 | 2246 | 3031
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of ethnicity information.
  Participants
    Race: American Indian or Alaska Native | 2 | 0 | 5 | 40 | 47
    Race: Asian | 20 | 25 | 88 | 313 | 446
    Race: Black | 21 | 23 | 149 | 611 | 804
    Race: Native Hawaiian or Pacific Islander | 1 | 0 | 11 | 29 | 41
    Race: White | 142 | 134 | 376 | 1915 | 2567
    Race: Not Permitted | 0 | 5 | 56 | 179 | 240
    Race: Other | 14 | 10 | 159 | 510 | 693
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Measure Description: Not Permitted means local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 47 | 38 | 328 | 1341 | 1754
    Ethnicity: Not Hispanic or Latino | 152 | 150 | 478 | 2123 | 2903
    Ethnicity: Not Permitted | 1 | 9 | 37 | 129 | 176
    Ethnicity: Missing | 0 | 0 | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 118 | 111 | 722 | 2927 | 3878
  Spain | 31 | 30 | 27 | 134 | 222
  Italy | 39 | 38 | 16 | 108 | 201
  United Kingdom | 0 | 0 | 33 | 144 | 177
  Sweden | 0 | 0 | 5 | 83 | 88
  Singapore | 1 | 8 | 7 | 44 | 60
  Switzerland | 0 | 0 | 13 | 44 | 57
  Netherlands | 0 | 0 | 2 | 45 | 47
  Germany | 3 | 1 | 12 | 27 | 43
  France | 0 | 0 | 2 | 25 | 27
  South Korea | 6 | 6 | 0 | 10 | 22
  Hong Kong | 2 | 2 | 2 | 0 | 6
  Japan | 0 | 0 | 1 | 4 | 5
  Taiwan | 0 | 1 | 2 | 2 | 5
Clinical Status (7-point ordinal scale) [Count of Participants; unit: Participants] — The 7-point ordinal scale is an assessment of the clinical status of participant at a given study day:1. Death;2.Hospitalized,on invasive mechanical ventilation or extracorporeal membrane oxygenation(ECMO);3.Hospitalized, on noninvasive ventilation or high-flow oxygen devices;4.Hospitalized,requiring low-flow supplemental oxygen;5.Hospitalized,not requiring supplemental oxygen - requiring ongoing medical care(COVID-19 related or otherwise);6.Hospitalized,not requiring supplemental oxygen - no longer requiring ongoing medical care(other than per-protocol RDV administration);7.Not hospitalized.
  Participants
    Score: 1 | 0 | 0 | 0 | 0 | 0
    Score: 2 | 4 | 9 | 844 | 0 | 857
    Score: 3 | 49 | 59 | 0 | 1069 | 1177
    Score: 4 | 113 | 108 | 0 | 2214 | 2435
    Score: 5 | 34 | 21 | 0 | 314 | 369
    Score: 6 | 0 | 0 | 0 | 0 | 0
    Score: 7 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants in Each Clinical Status Category as Assessed by a 7-Point Ordinal Scale on Day 14
Description: Clinical status was derived from death, hospital discharge, and the ordinal scale as follows: score of "1" was used for all days on or after the date of death; score of "7" was used for all days on or after discharged alive date; last assessment carried forward for any missing values.The scale is as follows: 1. Death; 2. Hospitalized, on invasive mechanical ventilation or ECMO; 3. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring low flow supplemental oxygen; 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6. Hospitalized, not requiring supplemental oxygen - no longer required ongoing medical care (other than per protocol remdesivir administration); 7. Not hospitalized. The odds ratio represents the odds of improvement in the ordinal scale for the Remdesivir for 10 days group vs the Remdesivir for 5 days group.
Time Frame: Day 14
Population: Full Analysis Set included participants who were randomized into part A of the study and received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Remdesivir (RDV) for 5 Days | Part A: Remdesivir for 10 Days
Number analyzed (Participants) | 200 | 197
percentage of participants
  Score: 1 | 8.0 | 10.7
  Score: 2 | 8.5 | 16.8
  Score: 3 | 4.0 | 5.1
  Score: 4 | 9.5 | 7.6
  Score: 5 | 6.0 | 6.1
  Score: 6 | 4.0 | 1.5
  Score: 7 | 60.0 | 52.3
Statistical Analysis 1: Comparison: Part A: Remdesivir (RDV) for 5 Days vs Part A: Remdesivir for 10 Days; Test type: Superiority; p = 0.1563, Proportional odds model — P-value was calculated using a proportional odds model with treatment as the independent variable and baseline clinical status as a continuous covariate; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.507 to 1.115]
Statistical Analysis 2: Comparison: Part A: Remdesivir (RDV) for 5 Days vs Part A: Remdesivir for 10 Days; Test type: Superiority; p = 0.0368, Proportional odds model — P-value was calculated using a proportional odds model with treatment as the independent variable; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.458 to 0.976]

2. Secondary Outcome: Part A: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent Adverse Events (TEAE) were defined as AEs with onset dates on or after the study treatment start date and no later than 30 days after the permanent discontinuation of the study treatment and/or the AEs that led to premature discontinuation of study treatment.
Time Frame: First dose date up to last dose date (maximum: 10 days) plus 30 days
Population: Part A: Safety Analysis Set included participants who were randomized into part A of the study and received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Remdesivir (RDV) for 5 Days | Part A: Remdesivir for 10 Days
Number analyzed (Participants) | 200 | 197
percentage of participants | 71.5 [64.7 to 77.6] | 75.1 [68.5 to 81.0]
Statistical Analysis 1: Comparison: Part A: Remdesivir (RDV) for 5 Days vs Part A: Remdesivir for 10 Days; Test type: Superiority; p = 0.7678, Cochran-Mantel-Haenszel — P-value for comparison of the percentages between the two groups was calculated using the Cochran-Mantel-Haenszel test stratified on baseline clinical status; Difference in Percentages = 1.3, 95% CI 2-sided [-7.4 to 10.0]

ADVERSE EVENTS:
Time Frame: Part A: First dose date up to the last dose date (maximum: 10 days) plus 30 days; Part B: First dose date up to the last dose date (maximum: 11 days) plus 30 days
Description: Part A: Safety Analysis Set included participants who were randomized into part A of the study and received at least 1 dose of study treatment;Part B: Expanded RDV-Treated Analysis Set included participants who were enrolled into part B of the study and received at least 1 dose of study treatment.
Arm/Group | Part A: Remdesivir (RDV) for 5 Days | Part A: Remdesivir for 10 Days | Part B: Remdesivir for 10 Days (Mechanically Ventilated Group) | Part B: Remdesivir for 10 Days (Extension Group)
All-Cause Mortality (participants affected / at risk) | 25/200 | 28/197 | 213/844 | 422/3597
Serious Adverse Events (participants affected / at risk) | 43/200 | 68/197 | 362/844 | 851/3597
Other Adverse Events (participants affected / at risk) | 79/200 | 92/197 | 508/844 | 1258/3597
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Remdesivir (RDV) for 5 Days (N=200) | Part A: Remdesivir for 10 Days (N=197) | Part B: Remdesivir for 10 Days (Mechanically Ventilated Group) (N=844) | Part B: Remdesivir for 10 Days (Extension Group) (N=3597)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 9
Bicytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 4 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 3 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 10 | 12
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 3
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 2 | 3
Cardiac arrest (Cardiac disorders) | 0 | 2 | 15 | 34
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 2 | 11
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 5
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 2 | 1
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 4
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 2 | 5
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 2 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 2 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0
Brain death (General disorders) | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 1 | 1
Death (General disorders) | 1 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 0 | 1 | 0
Hyperthermia malignant (General disorders) | 0 | 0 | 2 | 0
Multi-organ disorder (General disorders) | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 4 | 27 | 32
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pelvic mass (General disorders) | 0 | 0 | 0 | 1
Procedural failure (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 4 | 5
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 2 | 5
Cytokine storm (Immune system disorders) | 0 | 0 | 1 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 7 | 3
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Citrobacter bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 8 | 10 | 5 | 22
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 6 | 24
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 7 | 4
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 3 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 3 | 2 | 18 | 22
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 2 | 1 | 11 | 34
Septic shock (Infections and infestations) | 2 | 5 | 27 | 52
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Superinfection (Infections and infestations) | 0 | 0 | 1 | 1
Superinfection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Thrombophlebitis septic (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Viral myocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Viral sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Barotrauma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 4
Bacterial test positive (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 5 | 2
Blood pressure abnormal (Investigations) | 0 | 0 | 0 | 1
Coma scale abnormal (Investigations) | 0 | 0 | 0 | 1
Creatinine renal clearance abnormal (Investigations) | 0 | 0 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 2 | 4
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 1 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 2
Myocardial necrosis marker increased (Investigations) | 0 | 0 | 0 | 1
Oxygen consumption increased (Investigations) | 0 | 0 | 1 | 1
Oxygen saturation abnormal (Investigations) | 0 | 0 | 2 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 5
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 3 | 2 | 6 | 3
Troponin increased (Investigations) | 0 | 0 | 0 | 2
Urine output decreased (Investigations) | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 1
Brain injury (Nervous system disorders) | 0 | 0 | 3 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 3 | 4
Cerebral infarction (Nervous system disorders) | 0 | 0 | 2 | 3
Cerebral microhaemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 4 | 7
Coma (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 2
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 4 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Iiird nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 4
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 3
Seizure like phenomena (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 2 | 10
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 3 | 50 | 69
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 13 | 17
Renal impairment (Renal and urinary disorders) | 0 | 0 | 4 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Priapism (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 23 | 42
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 36 | 121
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 26
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Hyperoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 14 | 78
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6 | 25
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 9 | 32
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 22
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 14 | 71
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 59 | 254
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 4
Social stay hospitalisation (Social circumstances) | 0 | 0 | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 6 | 3
Distributive shock (Vascular disorders) | 0 | 0 | 0 | 3
Dry gangrene (Vascular disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Haemodynamic instability (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 3 | 23 | 53
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 3
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 1
Shock (Vascular disorders) | 0 | 0 | 7 | 11
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 2 | 4
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Remdesivir (RDV) for 5 Days (N=200) | Part A: Remdesivir for 10 Days (N=197) | Part B: Remdesivir for 10 Days (Mechanically Ventilated Group) (N=844) | Part B: Remdesivir for 10 Days (Extension Group) (N=3597)
Anaemia (Blood and lymphatic system disorders) | 7 | 7 | 88 | 104
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 47 | 42
Constipation (Gastrointestinal disorders) | 13 | 13 | 78 | 237
Diarrhoea (Gastrointestinal disorders) | 10 | 9 | 54 | 128
Nausea (Gastrointestinal disorders) | 20 | 17 | 28 | 220
Pyrexia (General disorders) | 9 | 3 | 65 | 101
Pneumonia (Infections and infestations) | 1 | 3 | 48 | 48
Alanine aminotransferase increased (Investigations) | 10 | 15 | 53 | 164
Aspartate aminotransferase increased (Investigations) | 8 | 13 | 66 | 126
Transaminases increased (Investigations) | 3 | 4 | 43 | 93
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 7 | 62 | 92
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 2 | 92 | 59
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 12 | 78 | 190
Agitation (Psychiatric disorders) | 2 | 4 | 74 | 47
Delirium (Psychiatric disorders) | 2 | 2 | 60 | 40
Insomnia (Psychiatric disorders) | 10 | 11 | 17 | 116
Acute kidney injury (Renal and urinary disorders) | 2 | 13 | 113 | 117
Deep vein thrombosis (Vascular disorders) | 4 | 5 | 50 | 55
Hypertension (Vascular disorders) | 5 | 6 | 92 | 67
Hypotension (Vascular disorders) | 8 | 9 | 99 | 166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2020-04-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT04292899/Prot_000.pdf
  • Statistical Analysis Plan: Part A (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04292899/SAP_001.pdf
  • Statistical Analysis Plan: Part B (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT04292899/SAP_002.pdf